CLINICAL TRIAL: NCT00630643
Title: A Phase I/IIa, Double-Blind, Placebo-Controlled, Dose-Escalation Study of NI-0401 in Patients With Moderate to Severe Active Crohn´s Disease
Brief Title: NI-0401 in Active Crohn's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Light Chain Bioscience - Novimmune SA (Industry)
Responsible Party: Dr Janeke Van der Woude, Erasmus Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NI-0401-01
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-02

CONDITIONS: Moderate to Severe Crohn's Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Biological: NI-0401 (anti-CD3 mAB)

INTERVENTIONS:
Biological: NI-0401 (anti-CD3 mAB) — 0.05 mg up to 10 mg
  Arms: 2
Drug: Placebo — Placebo
  Arms: 1

SUMMARY:
The purpose of the study is to assess the safety and tolerability of daily intravenous NI-0401 treatment, compared to matching placebo. And to assess the ability of NI-0401 to modulate the CD3 complex on T-cells.

ELIGIBILITY:
Main Inclusion Criteria:

1. Men and women between 18 and 70 years of age.
2. Crohn's Disease Activity Index (CDAI) between 220 and 450.
3. Raised plasma CRP level.
4. Endoscopic inflammation.
5. Crohn's disease of at least 6 months duration, with colitis, ileitis, or ileocolitis, confirmed by endoscopy and histology within 28 days of study day 1.

Main Exclusion criteria

1. Have received or are planned to receive immunization with a live vaccine within 6 weeks prior to receiving study drug and 12 weeks after treatment cessation.
2. Concomitant disease:

   * Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac, neurological or cerebral disease (including a history of seizure disorders or ongoing chronic active conditions such as chronic active hepatitis)
   * Previous diagnosis of, or known, malignancies
   * Severe infections, such as hepatitis, pneumonia or pyelonephritis, in the past three months. Less serious infections in the past 3 months, such as acute upper respiratory tract infection (colds) or uncompliant urinary tract infection are permitted at the discretion of the investigator
   * Active infection requiring antibiotic therapy
   * Serum anti HCV positive, serum HBsAg positive, serum anti-HIV positive
   * History of opportunistic infections such as herpes zoster within 2 months prior to screening, evidence of acute CMV or EBV, active Pneumocystic Carinii
   * History of active tuberculosis (TB) or currently undergoing treatment for TB. Patients with a positive TB skin test or chest x-ray are ineligible. Patients with a history of bacille Calmette Guerin (BCG) vaccination and a newly positive TB skin test or a chest X-ray showing fibrotic lesions consistent with previous TB are ineligible. The PPD skin test must be read between 48 and 72 hours
   * Stool examination positive for enteric pathogens, pathogenic ova or parasites, or Clostridium Difficile toxin within 4 weeks prior to Study Day 1

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of intravenous NI-0401 . | 24 weeks

SECONDARY OUTCOMES:
Immunological response defined as the percent change in the modulation of the CD3 complex on T-cells

CONTACTS AND LOCATIONS:
Overall Officials: Janeeke Van der Woude, MD, Principal Investigator — Erasmus Medisch Centrum